CLINICAL TRIAL: NCT06364839
Title: Liver Transplantation for Hepatocellular Carcinoma Arising in Non-cirrhotic Liver: a Propensity Score-matched Retrospective Cohort Study of Two National Databases
Status: Completed | Type: Observational
Sponsor: Xiao Xu (Other)
Responsible Party: Sponsor-Investigator, Xiao Xu, Principal Investigator, Clinical Professor,PHD,MD, Zhejiang University
Organization: Zhejiang University (Other)
Other Study IDs: CT2024-ZJU-OBS7
Record Dates: First submitted 2024-04-04; First posted 2024-04-15 (Actual); Last update posted 2024-04-15 (Actual); Status verified 2024-04

CONDITIONS: Hepatocellular Carcinoma, Non-cirrhotic Liver
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other:

SUMMARY:
Background: Majority of liver transplantation (LT) recipients for hepatocellular carcinoma (HCC) were concomitant with liver cirrhosis, while few researches focusing on recipients without cirrhosis. Here we aim to investigate the prognosis of non-cirrhosis HCC recipients, expecting to provide theoretical basis for further improvement of these patients.

Methods: This retrospective study analyze outcomes between adult HCC recipients arising in non-cirrhotic and cirrhotic liver from two national databases (CLTR and UNOS, January 2015 to December 2020). Based on important variables, 1:2 and 1:1 propensity score matching (PSM) were performed respectively.

ELIGIBILITY:
Inclusion Criteria:

* liver transplants, performed from January 2015 to December 2020

Exclusion Criteria:

* pediatric LT; LT for non-tumor lesions; LT for other malignant tumors (cholangiocarcinoma, carcinoma of gallbladder, mixed carcinoma, and secondary tumors); re-transplantation or combined liver-kidney transplantation; incomplete laboratory or clinical data; death within 1 week due to post-operative hemorrhage after LT.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Previously registered liver transplant recipients
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2024-02-20 (Actual); Primary Completion 2024-03-23 (Actual); Study Completion 2024-03-25 (Actual)

PRIMARY OUTCOMES:
Postoperative complications were evaluated by postoperative imaging and serological examination | 3 months
  Including rejection after liver transplantation, vascular complications, new metabolic diseases and so on
The overall survival rate was evaluated by follow-up investigation and outpatient review | 1-3 years
The tumor-free survival rate was evaluated by follow-up investigation and outpatient review | 1-3 years

CONTACTS AND LOCATIONS:
Locations (1):
- Xiao Xu, Hangzhou, Zhejiang, China